CLINICAL TRIAL: NCT06131801
Title: A Pharmacokinetic Study of Venetoclax Tablets Crushed and Dissolved Into a Solution in Children and Young Adults With Hematologic Malignancies
Brief Title: Pharmacokinetic Study of Venetoclax Tablets Crushed and Dissolved Into a Solution
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: Venetoclax PK
Record Dates: First submitted 2023-10-24; First posted 2023-11-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancy; Leukemia; Lymphoma; Acute Lymphocytic Leukemia; ALL; Acute Myelogenous Leukemia; AML; Chronic Myelogenous Leukemia; CML; Myeloproliferative Neoplasm; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Burkitt Lymphoma; T-cell Lymphoma; B Cell Lymphoma; Peripheral T Cell Lymphoma; Cutaneous B-Cell Lymphoma
Keywords: Venetoclax; Pediatric AML; Pediatric Relapsed/Refractory AML
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Burkitt Lymphoma; Lymphoma, T-Cell; Lymphoma, B-Cell; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (1-2 mL) collected from an existing venous or arterial access line. Patients < 14 kg (approximately 31 pounds) will be limited to 1 mL for each PK sample draw.
  OPTIONAL: An additional 3-4 mLs of cerebrospinal fluid (CSF) at any time point in which cerebrospinal fluid (CSF) is already being obtained as part of standard of care therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and Young Adults: Children and Young Adults who are prescribed venetoclax made from crushed tablets as part of their clinical care.
  Interventions: Other: 1. Drug: The Venetoclax PK study is collecting bodily fluid samples (ie., whole blood and optional cerebrospinal fluid) of patients prescribed venetoclax as crushed tablets per standard of care.

INTERVENTIONS:
Other: 1. Drug: The Venetoclax PK study is collecting bodily fluid samples (ie., whole blood and optional cerebrospinal fluid) of patients prescribed venetoclax as crushed tablets per standard of care. — Participants will receive Venetoclax as prescribed by their treating provider as part of their clinical care.

SUMMARY:
The use of venetoclax-based therapies for pediatric patients with relapsed or refractory malignancies is increasingly common outside of the clinical trial setting. For patients who cannot swallow tablets, it is common to crush the tablets and dissolve them in liquid to create a solution. However, no PK data exists in adults or children using crushed tablets dissolved in liquid in this manner, and as a result, the venetoclax exposure with this solution is unknown.

Primary Objectives

• To determine the pharmacokinetics of venetoclax when commercially available tablets are crushed and dissolved into a solution

Secondary Objectives

* To evaluate the safety of crushed venetoclax tablets administered as an oral solution
* To determine the pharmacokinetics of venetoclax solution in patients receiving concomitant strong and moderate CYP3A inhibitors
* To determine potential pharmacokinetic differences based on route of venetoclax solution administration (ie. PO vs NG tube vs G-tube)
* To determine the concentration of venetoclax in cerebral spinal fluid when administered as an oral solution

DETAILED DESCRIPTION:
Peripheral blood will be drawn at multiple time points to evaluate venetoclax pharmacokinetics in patients who are receiving venetoclax solution made from crushed tablets as part of their oncology treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be <39 years of age at time of study enrollment
* Diagnosis: Patients may have a diagnosis of any hematologic malignancy
* Central access: Patients must have an existing venous or arterial access line for PK blood draws
* Weight requirement: Patients must weigh at least 5.5 kg at the time of enrollment
* Venetoclax: Patients must be receiving any dose of venetoclax given as a solution made from crushed tablets by mouth (PO) or via nasogastric (NG), or G-tube as prescribed by their treating oncologist.
* Concurrent chemotherapy medications: Patients may receive venetoclax as a single agent or in combination with any other chemotherapeutic agents.

Exclusion Criteria:

* Pregnant women are excluded from this study because venetoclax has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued if the mother is treated with venetoclax.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on study treatment and for six months following completion.

Ages: 0 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients must be receiving any dose of venetoclax given as a solution made from crushed tablets by mouth (PO) or via nasogastric (NG), or G-tube as prescribed by their treating oncologist.
  Patients must be <39 years of age at time of study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: the observed peak plasma concentration (Cmax)
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: the time to peak (Tmax)
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: the apparent terminal phase elimination rate constant (β)
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: the terminal-phase elimination half-life (T1/2)
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: the areas under plasma concentration curve (AUC) over a 24-hour dose interval (AUC0-24) or for infinite time (AUC0-∞)
Clearance (CL) as measured by PK sampling (Peripheral Blood; Required) | Blood will be collected on one PK day between Days 5-12 after completion of the venetoclax dose ramp-up : within 1hr prior to the administration of venetoclax, then 2hrs, 5hrs, 12hrs, 18hrs and 24hrs after the administration of venetoclax.
  PK parameters of venetoclax will be described in peripheral blood including: oral clearance (CL/F) of venetoclax
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: the observed peak plasma concentration (Cmax)
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: the time to peak (Tmax)
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: the apparent terminal phase elimination rate constant (β)
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: the terminal-phase elimination half-life (T1/2)
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: the areas under plasma concentration curve (AUC) over a 24-hour dose interval (AUC0-24) or for infinite time (AUC0-∞)
Clearance (CL) as measured by PK sampling (Cerebrospinal Fluid; Optional) | Around Days 8, 15, 22, and/or 28, all +/- 3 days. Not all patients will have CSF collected at these time points.
  PK parameters of venetoclax will be described in cerebral spinal fluid including: oral clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Pommert, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin